CLINICAL TRIAL: NCT01475331
Title: The CHARM Trial: Chemotherapy for Ablation and Resolution of Mucinous Pancreatic Cysts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Matthew T. Moyer, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 33751
Record Dates: First submitted 2011-11-08; First posted 2011-11-21 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-02

CONDITIONS: Mucinous Pancreatic Cysts
Keywords: pancreatic cyst; chemotherapy; ethanol; ablation
MeSH Terms: conditions — Pancreatic Cyst | interventions — Ethanol; Saline Solution; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): Cyst will be lavaged for 3-5 minutes with Ethanol (alcohol 80%). Following lavage with Ethanol (alcohol 80%), The cyst will be infused with an admixture of chemotherapy drugs (Paclitaxel/ Gemcitabine) 3mg/ml paclitaxel and 19mg/ml gemcitabine.
  Interventions: Drug: Ethanol; Drug: Chemotherapy
- Study Group (Experimental): Cyst will be lavaged for 3-5 minutes with Normal Saline .. Following lavage with Normal Saline, The cyst will be infused with an admixture of chemotherapy drugs (Paclitaxel/ Gemcitabine) 3mg/ml paclitaxel and 19mg/ml gemcitabine.
  Interventions: Drug: Normal Saline; Drug: Chemotherapy

INTERVENTIONS:
Drug: Ethanol — Cysts will be lavaged for 3-5 minutes with 80% EtOH
  Arms: Control Group
Drug: Normal Saline — Cysts will be lavaged for 3-5 minutes with normal saline
  Arms: Study Group
Drug: Chemotherapy — Following lavage with either 80% ethanol (control group) or normal saline (study group), cysts will be injected with a cocktail of 3mg/ml paclitaxel and 19mg/ml gemcitabine.

SUMMARY:
The purpose of this study is to evaluate the efficacy of a chemotherapeutic cocktail with or without prior ethanol lavage for ablation of premalignant pancreatic cysts using endoscopic ultrasound-guided fine needle injection (EUS-FNI) for agent delivery.

DETAILED DESCRIPTION:
While about half of pancreatic cystic lesions have little to no malignant potential, mucinous cystic neoplasms (MCNs) and intraductal papillary mucinous neoplasms (IPMNs) carry a high potential for progression into pancreatic cancer. Therefore, either close radiographic surveillance or surgical resection is generally recommended for these cysts. However, pancreatic surgery is associated with a significant risk of morbidity and mortality and not all patients are good surgical candidates. As an alternative, endoscopic ultrasound-guided fine needle injection(EUS-FNI) has been shown to be moderately effective in ablating cystic lesions.

The goal of this investigation is to improve the efficacy and safety of this procedure when compared with previous versions of the technique. This study is designed to evaluate the efficacy of a chemotherapeutic cocktail with or without prior ethanol lavage for ablation of pancreatic cystic neoplasms using EUS-FNI for agent delivery. This paired, prospective, double-blind, randomized study will include 78 patients referred to the Penn State Hershey Medical Center. Mucinous or indeterminate pancreatic cysts of 1-5cm with less than 5 compartments and without clear communication with the main pancreatic duct will be included. Patients will be randomized in a 1:1 ratio into a control arm or study arm. Patients randomized to the control arm will receive ethanol lavage of the cyst followed by injection of two carefully selected chemotherapeutic agents. Study arm patients will receive a normal saline lavage followed by injection of the same chemotherapy admixture. Patients will be monitored for 2 hours post-procedure, and a follow-up CT will be performed at 6, and 12 months, or as determined necessary to evaluate cyst resolution. Patients may elect to undergo evaluation for surgical resection at any time, regardless of response, in which case a dedicated pathologist will evaluate any surgical specimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and older of any gender, ethnicity and race
* Voluntary enrollment and ability to give written informed consent
* Capable of safely undergoing endoscopy with deep sedation or general anesthesia
* Patients with previously-detected pancreatic cyst(s) 1-5 cm in diameter, including indeterminate cysts

Exclusion Criteria:

* Pancreatic cyst <1cm or >5cm
* Pancreatic cyst with clear communication with main pancreatic duct
* Clearly benign lesions by clinical and radiographic evaluation (pseudocysts and serous cystadenomas)
* Known or suspected pancreatic cancer or pathologic lymphadenopathy
* Septated cysts with > 5 compartments
* Coagulopathy (international normalized ratio > 1.6, platelets < 30,000)
* Evidence of active pancreatitis or pancreatic infection
* Patients having undergone endoscopic retrograde cholangiopancreatography (ERCP) within 72 hours
* Baseline lab values at the time of consent: white blood cells > 14 or < 2, hematocrit < 30, platelets < 30,000, INR > 1.6, abnormal CA19-9, lipase > 3 times the upper limit of normal, creatinine > 2.5, ALT > 210, total bilirubin > 2.5, positive qualitative beta-hCG.
* Any pre-existing or discovered medical condition that may, at the discretion of the investigator, interfere with the completion of and/or participation in the existing protocol.
* Pregnant, breastfeeding, or incarcerated individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Moyer MT, Sharzehi S, Mathew A, Levenick JM, Headlee BD, Blandford JT, Heisey HD, Birkholz JH, Ancrile BB, Maranki JL, Gusani NJ, McGarrity TJ, Dye CE. The Safety and Efficacy of an Alcohol-Free Pancreatic Cyst Ablation Protocol. Gastroenterology. 2017 Nov;153(5):1295-1303. doi: 10.1053/j.gastro.2017.08.009. Epub 2017 Aug 9. PMID 28802565

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Cyst will be lavaged for 3-5 minutes with Ethanol (alcohol 80%). Following lavage with Ethanol (alcohol 80%), The cyst will be infused with an admixture of(Paclitaxel/ Gemcitabine) 3mg/ml paclitaxel and 19mg/ml gemcitabine.
  Ethanol: Cysts will be lavaged for 3-5 minutes with 80% EtOH
  Chemotherapy: Following lavage with either 80% ethanol (control group) or normal saline (study group), cysts will be injected with a cocktail of 3mg/ml paclitaxel and 19mg/ml gemcitabine.
- Study Group: Cyst will be lavaged for 3-5 minutes with Normal Saline .. Following lavage with Normal Saline, The cyst will be infused with an admixture of(Paclitaxel/ Gemcitabine) 3mg/ml paclitaxel and 19mg/ml gemcitabine.
  Normal Saline: Cysts will be lavaged for 3-5 minutes with normal saline
  Chemotherapy: Following lavage with either 80% ethanol (control group) or normal saline (study group), cysts will be injected with a cocktail of 3mg/ml paclitaxel and 19mg/ml gemcitabine.
Period: Overall Study
Arm/Group | Control Group | Study Group
Started | 23 | 23
Completed | 18 | 21
Not Completed | 5 | 2
Not completed — Osteophyte obstruction of the proximal | 1 | 0
Not completed — excessive main duct communication | 1 | 1
Not completed — Loss of needle positioning due pt. cough | 1 | 0
Not completed — Sign of malignancy during the procedure | 2 | 0
Not completed — cyst found to be prohibitively small | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Study Group | Total
Number analyzed (Participants) | 18 | 21 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 8 | 12
  >=65 years | 14 | 13 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 5 | 11 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 16 | 19 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 21 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Changing in Cyst Volume
Description: The primary outcome of interest will be change in cyst size, as measured on initial, 6, and 12 month CT/MRI, or as determined necessary to evaluate cyst resolution. Cyst size was calculated by measuring x and y diameters and calculating cyst volume using the formula:4/3xpxr3 where r is the average of the cyst radius as measured on the initial, 6-month, and 12-month magnetic resonance imaging or computed tomography. Response was defined according to the same volume percentage reductions as described in previous trials where: complete response is a =>95% reduction in cyst volume, partial response is a 94%-75% reduction, and anon-response is <75% reduction in volume.11 The overall ablation rates in both arms were also compared with historical controls to assess the efficacy of the chemotherapeutic cocktail.
Time Frame: 6, and 12 months post procedure
Population: Intent to treat population (all participants at least one dose of intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 18 | 21
Participants
  Complete Response after 6 mon | 6 | 12
  Partial Response after 6 months | 5 | 4
  No Response after 6 months | 6 | 5
  Complete Response after 12 months | 11 | 14
  Partial Response after 12 months | 4 | 3
  No Response after 12 months | 3 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were determined and collected through study completion, an average of 1 year.
Arm/Group | Control Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/21
Other Adverse Events (participants affected / at risk) | 4/18 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=18) | Study Group (N=21)
acute pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — acute pancreatitis after ablation of 20-mm tail cyst requiring a 36- hour hospital stay
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=18) | Study Group (N=21)
abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0) — abdominal pain requiring unscheduled clinical evaluation and treatment for pain control

LIMITATIONS AND CAVEATS:
Because of small number of participants this single-center trial is still weakly powered to show these differences with high levels of scientific certainty.Study was limited to one ablation only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No